CLINICAL TRIAL: NCT03556982
Title: CD123-Targeted CAR-T in Treating Patients With Relapsed/Refractory Acute Myelocytic Leukemia（AML）
Brief Title: CART-123 FOR Relapsed/Refractory Acute Myelocytic Leukemia（AML）
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-123 FOR AML
Record Dates: First submitted 2018-06-03; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-03

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute Myeloid Leukemia; Relapsed; Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART-123 (Experimental): The relapsed/refractory AML patients will receive allogenic or autologous CD123-Targeted CAR-T cells infusion after FC chemotherapy.
  Interventions: Biological: CART-123 cells

INTERVENTIONS:
Biological: CART-123 cells — CD123-Targeted CAR-T cells are infused to patient received FC chemotherapy

SUMMARY:
The purpose of this study is to evaluate the safety and efficiency of CD123-Targeted CAR-T in Treating Patients with relapsed/refractory AML

DETAILED DESCRIPTION:
The relapsed/refractory AML patients will receive FC (F,Fludarabine，C，Cyclophosphamide) chemotherapy followed by infusion of allogenic or autologous CD123-Targeted CAR-T cells.No graft-versus-host disease (GVHD) prevention will be conducted before or after infusion. Dose-limiting toxicity,incidence of adverse events and disease response will be detected post-infusion.

ELIGIBILITY:
Inclusion Criteria:

* CD123-expressing AML must be assured and must be relapsed or refractory disease. According to current traditional therapies, there must be no available alternative curative therapies and subjects must be either ineligible for allogeneic stem cell transplant (SCT), have refused SCT, or have disease activity that prohibits SCT at this time.
* Estimated life expectancy ≥ 12 weeks (according to investigator's judgment)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* CD123 expression of the malignant cells must be detected by immunohistochemistry or by flow cytometry
* Patients must have measurable or evaluable disease at the time of enrollment, which may include any evidence of disease including minimal residual disease detected by flow cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis.
* Patients must have an healthy donor for T cells.
* Cardiac function: Left ventricular ejection fraction greater than or equal to 40% by MUGA or cardiac MRI, or fractional shortening greater than or equal to 28% by ECHO or left ventricular ejection fraction greater than or equal to 50% by ECHO.
* Renal function: Creatinine level of peripheral blood is required no greater than 133umol/L.
* Females of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects on the fetus.
* Patients with history of allogeneic stem cell transplantation are eligible if there is no evidence of active GVHD and no longer taking immunosuppressive agents for at least 30 days prior to enrollment.
* Ability to give informed consent.

Exclusion Criteria:

* Evident signs suggesting that patients are potentially allergic to cytokines.
* Frequent infection history and recent infection is uncontrolled.
* Patients with concomitant genetic syndrome: patients with Down syndrome, Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome.
* Active acute or chronic graft-versus-host disease (GVHD) or requirement of immunosuppressant medications for GVHD within 4 weeks of enrollment.
* Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary. For additional details regarding use of steroid and immunosuppressant medications.
* Pregnancy and nursing females.
* HIV infection.
* Active hepatitis B or active hepatitis C.
* Participation in a prior investigational study within 4 weeks prior to enrollment or longer if required by local regulation. Participation in non-therapeutic research studies is allowed.
* Patients with a known history or prior diagnosis of other serious immunologic, malignant or inflammatory disease.
* Other situations we think not eligible for participation in the research.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 28 days
Incidence of adverse events as assessed | 3 months
Disease response (CR or CRi) | 3 months

SECONDARY OUTCOMES:
Engraftment of transferred CD123+ CAR T cells | 28 days
CAR123-specific antibody level | 6 months
Duration of response | 1year
Progression Free Survival | 1year
Survival | 1year

CONTACTS AND LOCATIONS:
Overall Officials: HUISHENG AI, Study Chair — 307 Hospital of PLA
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing 100071, China

IPD SHARING:
Plan to Share IPD: Undecided